CLINICAL TRIAL: NCT06704568
Title: Respiratory-based Core Exercises in Early Postpartum Improve Abdominal Strength, Pulmonary Function, and Quality of Life
Brief Title: Core Exercise and Early Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emine Merve Ersever, Head of physiotherapy department of haymana vocational high school physiotherapy, Ankara University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-51381736-771
Record Dates: First submitted 2024-10-11; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Anxiety; Exercise Overtraining; Fatigue
Keywords: core stabilitation; fatigue; pospartum; breathing exercises
MeSH Terms: conditions — Overtraining Syndrome; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1st group N=30 control group, 2nd group N=30 core exercise group, 3rd group N=30 breathing exercises group will be randomly divided into 3 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core exercise and early pospartum (Experimental): Unlike the control group; core exercises for 20-30 minutes, 3 days a week for 8 weeks, and respiratory exercises combined with core exercises for the respiratory exercises group
  Interventions: Other: exercise
- breathing exercise (Experimental): Slow and controlled breathing exercises will be performed starting with 5 seconds of inhalation and 5 seconds of exhalation twice a day for 10 minutes, 5 days a week for eight weeks, with a 10-second diaphragmatic breathing cycle (6 breaths/minute). The finger counting method will be recommended so that participants can easily follow the 5-second inhalation and 5-second exhalation cycles. The exercises can be done sitting or lying down. The individuals will be taught the differences between the two by switching between normal and deep breathing a few times. The respiratory exercises will be finished with relaxation exercises.
  Interventions: Other: exercise
- control (Experimental): No application will be made to the control group.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Unlike the control group; core exercises for 20-30 minutes, 3 days a week for 8 weeks, and respiratory exercises combined with core exercises for the respiratory exercises group: Slow and controlled breathing exercises will be performed starting with 5 seconds of inhalation and 5 seconds of exhalation twice a day for 10 minutes, 5 days a week for eight weeks, with a 10-second diaphragmatic breathing cycle (6 breaths/minute). The finger counting method will be recommended so that participants can easily follow the 5-second inhalation and 5-second exhalation cycles. The exercises can be done sitting or lying down. The individuals will be taught the differences between the two by switching between normal and deep breathing a few times. The respiratory exercises will be finished with relaxation exercises.

SUMMARY:
This study aimed to investigate the positive effects of abdominal core exercises and deep breathing exercises on abdominal muscle strength, pulmonary function, fatigue, and quality of life in the early postnatal period (1-6 months).

DETAILED DESCRIPTION:
The study will include 90 women who meet the inclusion criteria. Considering α < 0.05 and β = 0.2 (standard values that allow 90% power in sample size calculations), 3 groups of 30 participants were determined by considering at least 25 participants for each group based on an estimated 20% probability of loss during follow-up. 3 groups will be randomized as 1st group N=30 control group, 2nd group N=30 core exercise group, 3rd group N=30 respiratory exercises group. Unlike the control group; core exercises for 20 min-30 min 3 days a week for 8 weeks, respiratory exercises combined with core exercises for the respiratory exercises group: Starting with slow and controlled breathing exercises, it will be performed twice a day, 5 days a week for 8 weeks, 10 minutes, 5 seconds inhalation and 5 seconds exhalation, with a 10-second diaphragmatic breathing cycle (6 breaths/minute). The finger counting method will be recommended so that participants can easily follow the 5-second inhale and 5-second exhale cycles. The exercises can be done sitting or lying down. The individuals will be taught the differences between the two by switching between normal and deep breaths several times. The breathing exercises will be finished with relaxation exercises. The researchers created the core stabilization exercise program based on previous studies conducted by Litos (2014) and Horsley (2020) and in compliance with the guidelines of the Association of Obstetricians and Gynecologists (ACOG). The socio-demographic information and clinical characteristics of the participants in all three groups who meet the inclusion criteria and voluntarily agree to participate in the study will be questioned with the 'postpartum follow-up form'. Core endurance tests, respiratory tests, and fatigue assessments will be evaluated before and after the 8-week exercise and recorded on the form. For core measurement, three basic endurance tests will be performed, namely the trunk flexor endurance test and bilateral side bridge tests, following the Trunk Muscle Endurance Test protocol recommended by McGill et al. All movements will be performed after sufficient practice and the participants will be expected to try to maintain a static posture for as long as possible. Participants will be seated with their knees bent at 90◦ for the trunk flexor endurance test and their feet will be fixed. Then, participants will lean on the 60-degree trunk support with their hands clasped in front of their chests. Then, the trunk support will be pulled back 3 cm and they will be asked to maintain this posture for as long as possible. The test will be stopped when the participants lose their posture or their backs touch the support. Bilateral side bridge tests involve participants lying on their sides and lifting their trunks with their knees straight. One foot is placed in front of the other, hips are lifted and they will support their weight only with their elbows. The test will be stopped when the side-lying posture is lost or their hips drop to the mat. Respiratory tests will be performed with an analog spirometer. The maternal quality of life, and maternal perceived quality of life (MAPP-QOL) questionnaire was developed by Hill et al. (2006) and is based on the Quality of Life Index (QLI) of Ferrans et al. (1998). This questionnaire consists of thirty-eight items divided into five subcategories: Psychological/Baby (8 items), Socioeconomic (9 items), Relational/Partner (4 items), Relational/Family-Friends (9 items), and Health and Functioning (8 items). The internal consistency reliability (Cronbach's alpha) of the maternal quality of life questionnaire is R = 0.96 and the test and retest reliability at two-week intervals is R = 0.74. The level of fatigue perceived by individuals during the postpartum period will be recorded using the "Borg Fatigue Scale". Individuals will be asked to evaluate the level of fatigue they feel between 0 and 10. Individuals will be video-called at 2-week intervals to check their exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Having given birth within the last 1-6 months
2. Being between the ages of 18-45
3. Having a singleton pregnancy
4. Willingness to participate in the study
5. No history of physical or mental illness.

Exclusion Criteria:

1. Those with postpartum anemia
2. Those with postpartum respiratory tract infections
3. Those whose newborns were hospitalized for any reason
4. Those who gave birth to multiple babies
5. Those with a history of chronic back pain
6. Those with neurological symptoms
7. Those with cardiovascular and respiratory problems

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Having given birth within the last 1-6 months
Enrollment: 90 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Static Trunk Endurance Test | 8 week
  For endurance measurement,three core endurance tests were performed following the protocol of the TEMT. the trunk flexor endurance test and the bilateral side bridge tests. All movements were conducted after sufficient practice to eliminate any bias towards cognition, and the subjects aimed to maintain a static posture for as long as possible. The subjects sat with knees bent at 90° on the table for the trunk flexor endurance test, and their feet were held in place by a belt. Afterwards, they crossed their hands in front of their chests, leaned against the 60 degree trunk support, pulled the trunk support back 3 cm, and maintained this posture for as long as possible.The examination was stopped when the posture of lying on their side was lost or when their buttocks fell to the mat

SECONDARY OUTCOMES:
quality of life test | 8 week
  The second outcome measure was the quality of life and controlling factors and fatique Participants' postpartum quality of life was evaluated with the Maternal Postpartum Quality of Life (MAPPQOL) [16]. Postpartum quality of life is a scale that is evaluated according to the perception of the mother and consists of five sub-dimensions and a total of 40 items. Sub-dimensions of the scale; kinship consists of family friend (nine items), socioeconomic (nine items), spouse (five items), health (eight items), and psychological (nine items) dimensions. The scale assesses how satisfied and important mothers feel at four to six weeks post discharge postpartum. The scale consists of two parts. In the first part, satisfaction with each item is questioned, and in the second part, the importance is questioned.
Pulmonary Function Test | 8 week
  Pulmonary function test was done using a portable machine-a spirometer by COSMED technologies, USA. Variables that were used for this study included the following -forced vital capacity (L), forced expiratory volume in the first second (L), peak expiratory flow rate (L/s), and three tests were taken. The best value was entered in the datasheet

CONTACTS AND LOCATIONS:
Locations (1):
- Haymana State Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 mount

REFERENCES:
- [Background] Kim S, Yi D, Yim J. The Effect of Core Exercise Using Online Videoconferencing Platform and Offline-Based Intervention in Postpartum Woman with Diastasis Recti Abdominis. Int J Environ Res Public Health. 2022 Jun 8;19(12):7031. doi: 10.3390/ijerph19127031. PMID 35742279